CLINICAL TRIAL: NCT04208321
Title: A Phase 1, First-In-Human, Randomized, Double-Blind, Placebo-Controlled, Single Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of Single Oral Doses of VT-1598 in Healthy Adult Subjects
Brief Title: Safety and Pharmacokinetics of VT-1598
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0087; HHSN272201500007I
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Results first posted 2023-01-11 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2020-01-31

CONDITIONS: Coccidioidomycosis
Keywords: Adults; Healthy; Pharmacokinetics; Phase 1; Safety; Single Oral Doses; Tolerability; VT-1598
MeSH Terms: conditions — Coccidioidomycosis | interventions — VT-1598

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1 (Experimental): 40 mg (1 tablet of 40 mg) of VT-1598 administered orally as a single dose, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), while fasting on Day 1 in a double-blind manner.
  Interventions: Other: Placebo; Drug: VT-1598
- Cohort 2 (Experimental): 80 mg (2 tablets of 40 mg) of VT-1598 administered orally as a single dose, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), while fasting on Day 1 in a double-blind manner.
  Interventions: Other: Placebo; Drug: VT-1598
- Cohort 3 (Experimental): 160 mg (4 tablets of 40 mg) of VT-1598 administered orally as a single dose, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), while fasting on Day 1 in a double-blind manner.
  Interventions: Other: Placebo; Drug: VT-1598
- Cohort 4 (Experimental): 320 mg (4 tablets of 80 mg) of VT-1598 administered orally as a single dose, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), while fasting on Day 1 in a double-blind manner.
  Interventions: Other: Placebo; Drug: VT-1598
- Cohort 5 (Experimental): 640 mg (8 tablets of 80 mg) of VT-1598 administered orally as a single dose, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), while fasting on Day 1 in a double-blind manner.
  Interventions: Other: Placebo; Drug: VT-1598
- Cohort 6 (Experimental): 160 mg (4 tablets of 40 mg) of VT-1598 administered orally as a single dose, n=6, or matching placebo, n=2, after high-calorie, high-fat meal on Day 1 in a double-blind manner.
  Interventions: Other: Placebo; Drug: VT-1598

INTERVENTIONS:
Other: Placebo — Placebo will be supplied as matching tablets (to 40 mg and 80 mg VT-1598 tablets) containing the inactive components of VT-1598.
Drug: VT-1598 — VT-1598 is a novel oral agent for the treatment of fungal infections. It will be supplied as 40 mg and 80 mg tablets.

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose study in healthy adult subjects ages 18 - 45 years inclusive. It is designed to evaluate the safety and PK of single oral doses of VT-1598. Forty-eight subjects will be enrolled in the study at 1 site in the US and randomized to receive either VT-1598 or placebo in 6 dosage cohorts (five fasted cohorts and one fed cohort). Each cohort will have 8 subjects; 6 subjects will receive a single oral dose of VT-1598 and 2 subjects will receive matching placebo. Cohorts 1 - 5 will include 2 sentinel subjects randomized to different treatments. Cohort 6 (receiving treatment after being fed a high-calorie, high-fat meal) will not include sentinel subjects. Subjects will be admitted to the study site before dosing and remain at the study site for safety monitoring and PK assessments for at least 72 hours post-dose. Subjects will return to the study site on study Days 7, 14, and 21 for outpatient safety monitoring and PK assessments. There are no formal hypotheses being tested in this Phase 1 trial study. The primary objectives of this study are 1) to determine the safety of single-ascending oral doses of VT-1598 in healthy adult subjects in a fasted state, and 2) to determine the safety of single oral dose of VT-1598 in healthy adult subjects in a fed state.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose study in healthy adult subjects ages 18 - 45 years inclusive. It is designed to evaluate the safety and PK of single oral doses of VT-1598. Forty-eight subjects will be enrolled in the study at 1 site in the US and randomized to receive either VT-1598 or placebo in 6 dosage cohorts (five fasted cohorts and one fed cohort). Cohorts 1 - 4 will run sequentially, but Cohorts 5 and 6 may be started concurrently. Each cohort will have 8 subjects; 6 subjects will receive a single oral dose of VT-1598 and 2 subjects will receive matching placebo. Cohorts 1 - 5 will include 2 sentinel subjects randomized to different treatments. Cohort 6 (receiving treatment after being fed a high-calorie, high-fat meal) will not include sentinel subjects. VT-1598 will be administered in the following escalation schedule: Cohort 1 will receive 40 mg dose, Cohort 2 will receive 80 mg dose, Cohort 3 will receive 160 mg dose, Cohort 4 will receive 320 mg dose, Cohort 5 will receive 640 mg dose, and Cohort 6 (fed cohort) will receive 160 mg dose. Subjects will be admitted to the study site before dosing and remain at the study site for safety monitoring and PK assessments for at least 72 hours post-dose. Subjects will return to the study site on study Days 7, 14, and 21 for outpatient safety monitoring and PK assessments. There are no formal hypotheses being tested in this Phase 1 trial study. The primary objectives of this study are 1) to determine the safety of single-ascending oral doses of VT-1598 in healthy adult subjects in a fasted state, and 2) to determine the safety of single oral dose of VT-1598 in healthy adult subjects in a fed state. The secondary objectives of this study are 1) to determine the pharmacokinetic (PK) profile in plasma and urine of VT-1598 and its primary metabolite, VT-11134, in healthy adult subjects, and 2) to determine the effect of a high-fat, high-calorie meal on the PK profile of VT-1598 and VT-11134 when a single oral dose of VT-1598 is given.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent and authorization for use of protected health information.
2. Willing and able to comply with protocol requirements, instructions, and protocol-stated restrictions (including confinement to the Clinical Research Unit (CRU)) and is likely to complete the study as planned.
3. Male or female subjects, 18 - 45 years of age (inclusive).
4. Subject is in good health to be safely enrolled in this protocol as determined by medical history and physical exam.
5. Body Mass Index (BMI) of 18 - 35 kg / m^2, inclusive, and minimum weight of 50 kg.
6. If a female participant is of childbearing potential*, she must use a highly effective contraceptive method** from 30 days before enrollment through the 3 months after dosing.

   *A woman is considered of childbearing potential unless post-menopausal (subject is at least 50 years old and has history of >/=2 years without menses without other known or suspected cause and has a Follicle Stimulating Hormone (FSH) level >40 IU/L), or permanently surgically sterilized.

   **A highly effective contraceptive method includes surgical sterilization methods such as tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful tubal obliteration (e.g., Essure(R)) with documented radiological confirmation test at least 90 days after the procedure, or long-acting reversible contraception (progestin-releasing subdermal implants, copper intrauterine devices (IUDs), levonorgesterel-releasing IUDs).
7. Males* having sexual intercourse with women of childbearing potential must agree to consistent use of condoms from study product administration through 3 months after dosing**.

   *Including vasectomized men.

   **And must also agree to not donate sperm during the same time period.
8. Subject has adequate venous access for blood collection.

Exclusion Criteria:

1. Has a chronic condition that may increase risk to subject or interfere with endpoint assessment (e.g., liver disease, kidney disease, immunodeficiency).
2. Chronic condition diagnosed within 90 days of the screening visit.
3. Unstable chronic disease* within 6 months of the screening visit.

   *As defined by need for medical intervention that lead to a change in medications and/or required hospitalization, surgery/procedure, or ED/urgent care visit
4. History of psychiatric condition that has required hospitalization in the last 5 years or patient is considered unstable by study investigator.
5. Any condition that in the opinion of the Investigator could significantly impact drug absorption, distribution, or elimination.
6. Any out of normal range laboratory value* at screening or enrollment.

   *A laboratory value that is Grade 1 (with the exception of alanine aminotransferase (ALT), aspartate aminotransferase (AST), Total bilirubin, hemoglobin or serum creatinine) will be allowed if not considered to be clinically significant by the investigator.
7. Abnormal Electrocardiograms (ECGs).
8. Electrocardiographic QTcF interval >430 msec for males and >450 msec for females at Screening.
9. Positive test for antibodies to Human Immunodeficiency Virus-1 (HIV-1), Human Immunodeficiency Virus-2 (HIV-2), Hepatitis B surface antigen (HBsAg), or Hepatitis C (HCV).
10. Positive urine drug test. The drugs that will be screened for includes amphetamines, barbiturates , cocaine, opiates, cannabinoids, phencyclidine, and benzodiazepines.
11. Female subject of childbearing potential who is pregnant*, lactating, or planning to become pregnant during the study period or 3 months after the final dose of study product.

    *Having a positive serum pregnancy test at the Screening Visit or any other specified time point prior to the dose of study product.
12. Received any study product in a clinical trial within 30 days prior to Screening.
13. Admitted or documented illicit drug use or alcohol abuse within 6 months prior to Screening or during their participation in the trial.
14. Consumed alcohol within 72 hours of Day -1, until after the visit to the Clinical Research Unit (CRU) on Day 14 or have a positive alcohol test at Screening or on admission to the CRU.
15. Tobacco* use within 90 days prior to the Screening Visit or while a subject is enrolled in the study or a positive urine drug test for cotinine.

    *Tobacco use includes vaping, smoking tobacco, the use of snuff and chewing tobacco, and other nicotine or nicotine- containing products
16. Use of prescription drugs within 14 days prior to the dose of study product with the exception of hormonal contraceptives, which are permitted throughout the study.
17. Received any non-prescription medications, vitamins, or dietary supplements* within 7 days of dosing, unless prior approval is granted by both the Investigator and the Sponsor.

    *Excluded from this list is intermittent use of acetaminophen at doses of < / = 2 g / day or ibuprofen < / = 1200 mg / day. Herbal supplements must be discontinued 7 days prior to the dose of the study product.
18. History of intolerance or hypersensitivity to azole antifungals.
19. Blood donation or other significant blood loss within 60 days of screening and for the duration of the study.
20. Inability or difficulty swallowing whole capsules/tablets and/or multiple capsules/tablets.
21. Consumption of beverages and foods containing caffeine for 24 hours prior to Day -1 until discharge from the CRU on Day 4.
22. Consumption of grapefruit, or juices containing grapefruit or Seville oranges within 7 days prior to the scheduled dose of the study product until after the visit to the CRU on Day 14.
23. Subject has plans to enroll or is already enrolled in another clinical trial that could interfere with safety assessment of the investigational product at any time during the study period*.

    *Includes trials that have a study intervention such as a drug, biologic, or device
24. Having dietary restrictions that would preclude the subject from participating in either fed or fasting cohorts.
25. Having sensitivity or allergy to aspirin.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Early Phase Services Clinical Research Unit, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants included healthy adult male and female subjects aged 18-45 (inclusive). Participants were recruited from the local community to ensure that male, female, and minorities (African American, Native American, Asian, and Hispanics) were represented in the enrolled population. Participants were enrolled between 29SEP2020 and 17NOV2021.
Groups:
- 40 mg Fasted: 40 mg (1 tablet of 40 mg) of VT-1598 administered orally as a single dose, while fasting on Day 1 in a double-blind manner.
  VT-1598: VT-1598 is a novel oral agent for the treatment of fungal infections. It is supplied as 40 mg and 80 mg tablets.
- 80 mg Fasted: 80 mg (2 tablets of 40 mg) of VT-1598 administered orally as a single dose, while fasting on Day 1 in a double-blind manner.
  VT-1598: VT-1598 is a novel oral agent for the treatment of fungal infections. It is supplied as 40 mg and 80 mg tablets.
- 160 mg Fasted: 160 mg (4 tablets of 40 mg) of VT-1598 administered orally as a single dose, while fasting on Day 1 in a double-blind manner.
  VT-1598: VT-1598 is a novel oral agent for the treatment of fungal infections. It is supplied as 40 mg and 80 mg tablets.
- 160 mg Fed: 160 mg (4 tablets of 40 mg) of VT-1598 administered orally as a single dose, after a high-calorie, high-fat meal on Day 1 in a double-blind manner.
  VT-1598: VT-1598 is a novel oral agent for the treatment of fungal infections. It is supplied as 40 mg and 80 mg tablets.
- 320 mg Fasted: 320 mg (4 tablets of 80 mg) of VT-1598 administered orally as a single dose, while fasting on Day 1 in a double-blind manner.
  VT-1598: VT-1598 is a novel oral agent for the treatment of fungal infections. It is supplied as 40 mg and 80 mg tablets.
- 640 mg Fasted: 640 mg (8 tablets of 80 mg) of VT-1598 administered orally as a single dose, while fasting on Day 1 in a double-blind manner.
  VT-1598: VT-1598 is a novel oral agent for the treatment of fungal infections. It is supplied as 40 mg and 80 mg tablets.
- Placebo: Placebo participants across all cohorts: 40 mg (1 tablet of 40 mg) while fasting on Day 1; 80 mg (2 tablets of 40 mg) while fasting on Day 1; 160 mg (4 tablets of 40 mg) while fasting on Day 1; 160 mg (4 tablets of 40 mg) after a high-calorie, high-fat meal on Day 1; 320 mg (4 tablets of 80 mg) while fasting on Day 1; or 640 mg (8 tablets of 80 mg) while fasting on Day 1 of matching placebo administered orally as a single dose in a double-blind manner.
  Placebo: Placebo is supplied in matching tablets (to 40 mg and 80 mg VT-1598 tablets) containing the inactive components of VT-1598.
Period: Overall Study
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 12
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes the number of participants randomized.
Groups:
- 40 mg Fasted: 40 mg of VT-1598 administered orally as a single dose, while fasting on Day 1 in a double-blind manner.
- 80 mg Fasted: 80 mg of VT-1598 administered orally as a single dose, while fasting on Day 1 in a double-blind manner.
- 160 mg Fasted: 160 mg of VT-1598 administered orally as a single dose, while fasting on Day 1 in a double-blind manner.
- 160 mg Fed: 160 mg of VT-1598 administered orally as a single dose, after a high-calorie, high-fat meal on Day 1 in a double-blind manner.
- 320 mg Fasted: 320 mg of VT-1598 administered orally as a single dose, while fasting on Day 1 in a double-blind manner.
- 640 mg Fasted: 640 mg of VT-1598 administered orally as a single dose, while fasting on Day 1 in a double-blind manner.
- Placebo: Placebo participants across all cohorts given matching placebo administered orally as a single dose in a double-blind manner.
- Total: Total of all reporting groups
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (6.4) | 33.8 (5.2) | 34.5 (2.4) | 39.5 (3.4) | 38.3 (8.9) | 38.3 (6.3) | 33.3 (6.1) | 35.5 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 3 | 3 | 2 | 4 | 20
  Male | 4 | 4 | 2 | 3 | 3 | 4 | 8 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 3 | 4 | 3 | 4 | 6 | 27
  Not Hispanic or Latino | 2 | 3 | 3 | 2 | 3 | 1 | 5 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 1 | 2 | 1 | 4 | 15
  White | 4 | 4 | 3 | 5 | 4 | 5 | 8 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 163.23 (5.51) | 169.62 (11.32) | 163.63 (8.47) | 170.75 (13.51) | 166.05 (14.13) | 168.33 (11.65) | 174.16 (12.14) | 168.74 (11.42)
Weight [Mean (Standard Deviation); unit: kg] | 70.28 (15.26) | 90.08 (21.19) | 72.70 (6.88) | 77.77 (16.98) | 80.32 (18.76) | 84.42 (12.74) | 88.41 (14.76) | 81.55 (16.26)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.17 (4.23) | 30.83 (4.16) | 27.18 (2.38) | 26.47 (3.09) | 28.95 (4.28) | 30.05 (5.11) | 29.07 (3.10) | 28.47 (3.86)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Adverse events (AEs) are defined as any untoward medical occurrence regardless of its causal relationship to study treatment. Number of participants with an AE are summarized by MedDRA System Organ Class (SOC). Each subject was counted once per SOC. If a condition was present at screening, it was not considered an AE unless the severity worsened.
Time Frame: Day 1 through Day 21
Population: Safety Population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants
  General disorders and administration site conditions | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Infections and infestations | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Injury, poisoning and procedural complications | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Investigations | 6 | 6 | 6 | 5 | 3 | 5 | 11
  Musculoskeletal and connective tissue disorders | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Nervous system disorders | 0 | 0 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Abnormal Chemistry Laboratory Toxicity Results
Description: Laboratory parameters and associated thresholds include albumin <=3.4 g/dL, glucose <= 69 mg/dL or >=106 mg/dL, blood urea nitrogen (BUN) >= 21 mg/dL, potassium >=5.2 mEq/L or <=3.4 mEq/L, calcium < 8.7 mg/dL or >=10.3 mg/dL, sodium <=132 mEq/L or >=144 mEq/L, total protein <=5.9 g/dL, creatinine >=1.3 mg/dL (male) or >= 1.0 mg/dL (female), creatine phosphokinase >= 308 U/L (male) or >=192 U/L (female), phosphorus <=2.4 mg/dL, alkaline phosphatase >= 130 IU/L (males) or >= 105 IU/L (female), aspartate aminotransferase >= 39.9 U/L (male) or >= 31.9 U/L (female), alanine aminotransferase >=40.9 U/L (male) or >= 32.9 U/L (female), total bilirubin >=1.2 mg/dL, direct bilirubin >=0.2 mg/dL, magnesium <=1.6 mg/dL, and serum cortisol <= 4 ug/dL. If a clinical chemistry laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Baseline (Day -1) through Day 21
Population: Safety Population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants
  Albumin, Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, Increase | 4 | 2 | 3 | 3 | 1 | 3 | 4
  Blood Urea Nitrogen, Increase | 1 | 0 | 1 | 0 | 0 | 1 | 1
  Potassium, Decrease | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Potassium, Increase | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Calcium, Decrease | 0 | 1 | 0 | 1 | 2 | 0 | 3
  Calcium, Increase | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Sodium, Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Sodium, Increase | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Total Protein, Decrease | 1 | 1 | 1 | 0 | 0 | 0 | 3
  Creatinine, Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatine Phosphokinase, Increase | 2 | 0 | 2 | 0 | 0 | 2 | 4
  Phosphorus, Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase, Increase | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase, Increase | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Alanine Aminotransferase, Increase | 0 | 1 | 1 | 1 | 0 | 0 | 1
  Total Bilirubin, Increase | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Magnesium, Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serum Cortisol, Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 2

3. Primary Outcome: Number of Participants With Abnormal Hematology Laboratory Toxicity Results
Description: Laboratory parameters and associated thresholds for adverse events include hemoglobin <= 12.2 g/dL (male) or <= 10.8 g/dL (female), hematocrit <= 36.1 % (male) or <= 32.6 % (female), lymphocyte count <= 799 cell/mm3, neutrophil count <= 1,299 cell/mm3 (African Americans) or <= 1,699 cell/mm3 (all others), monocyte count >= 1001 cell/mm3, eosinophil count >= 871 cell/mm3, basophil count >= 101 cell/mm3, platelet count <= 150 x 10^3/mm3, red blood cell (RBC) count <= 4.1 x 10^6/uL (male) or <= 3.7 x 10^6/uL (female), and white blood cell (WBC) count >= 9,001 cell/mm3 or <= 2,499 cell/mm3 (African American Males) or >= 11,001 cell/mm3 or <= 2,499 cell/mm3 (African American Females) or >= 10,001 cell/mm3 or <= 3,999 cell/mm3 (all others). If a result met the threshold for an AE at baseline, subsequent results were only considered to be an AE if the grading worsened in severity.
Time Frame: Baseline (Day -1) through Day 21
Population: Safety Population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants
  Hemoglobin, Decrease | 1 | 1 | 0 | 0 | 0 | 0 | 1
  Hematocrit, Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, Decrease | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophils, Decrease | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Monocytes, Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils, Increase | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Basophils, Increase | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Platelets, Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Red Blood Cell, Decrease | 1 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell, Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White Blood Cell, Increase | 0 | 1 | 0 | 0 | 0 | 0 | 1

4. Primary Outcome: Number of Participants With Abnormal Coagulation Laboratory Toxicity Results
Description: Laboratory parameters include prothrombin time (PT), activated partial prothrombin time (PTT), and prothrombin international normalized ratio (INR). Thresholds for adverse events were considered as PT >= 11.6 s, PTT >= 30.1 s, INR >= 1.2. If a coagulation laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Baseline (Day -1) through Day 21
Population: Safety Population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants
  Activated Partial Thromboplastin Time, Increase | 0 | 0 | 1 | 2 | 0 | 1 | 2
  Prothrombin Time, Increase | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Prothrombin International Normalized Ratio, Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Urinalysis Laboratory Toxicity Results
Description: The only graded urinalysis laboratory parameter was red blood cells (RBC) by complete urinalysis. The threshold for adverse events was considered as >=3. If a urinalysis laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Baseline (Day -1) through Day 21
Population: Safety Population: All participants that received any amount of study product with complete urinalysis test performed.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted | Placebo
Number analyzed (Participants) | 2 | 3 | 4 | 4 | 3 | 3 | 3
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 2

6. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Toxicity Results
Description: Each participant is only counted once per toxicity grade for the worst severity recorded. The only ECG parameter graded was QTcF interval with a threshold of >= 30 msec. If an ECG value met the threshold for an AE at baseline, subsequent safety ECG results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 1 through Day 21
Population: Safety Population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Vital Signs
Description: Each participant is only counted once per toxicity grade for the worst severity recorded. Vital sign parameters include systolic blood pressure (BP), diastolic BP, pulse, respiratory rate, and temperature. Thresholds for abnormal vital signs were considered as systolic BP >= 141 mmHg or <= 89 mmHg, diastolic BP >= 91 mmHg, pulse <= 54 bpm (baseline > 60 bpm) or <=50 (baseline <= 60 bpm) or >= 101 bpm, respiratory rate >= 17 breaths per minute, and temperature >= 38.0 degrees Celsius. If a vital sign result met the threshold for an AE at baseline, subsequent vital sign results were only considered to be an AE if the grading worsened in severity.
Time Frame: Baseline (Day -1) through Day 21
Population: Safety Population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants
  Systolic Blood Pressure, Decrease | 2 | 1 | 0 | 0 | 0 | 0 | 1
  Systolic Blood Pressure, Increase | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Diastolic Blood Pressure, Increase | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse, Decrease | 1 | 2 | 2 | 1 | 0 | 1 | 2
  Pulse, Increase | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory Rate, Increase | 4 | 5 | 5 | 2 | 4 | 2 | 6
  Temperature, Increase | 0 | 1 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: VT-1598 Concentrations in Plasma
Description: Mean and standard deviation of VT-1598 concentrations in plasma by nominal time point.
Time Frame: 0 hours (h), 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 14 h, 24 h, 36 h, 48 h, 60 h, 72 h, 144 h, 312 h, and 480 h post dose
Population: PK Analysis Subset: all participants who received VT-1598 and have at least 1 quantifiable post dose plasma or urine sample with measurable drug or metabolite concentration, as well as no protocol deviations that would likely affect pharmacokinetic (PK) results and who have an evaluable plasma or urine concentration for either VT-1598 or VT-11134 from which at least a subset of the designated PK parameters can be determined.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL
  0 h | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  0.5 h | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  1 h | 0.000 (0.000) | 0.000 (0.000) | 6.417 (9.941) | 4.333 (6.780) | 8.117 (12.574) | 18.983 (24.670)
  1.5 h | 4.733 (7.642) | 7.067 (11.546) | 19.317 (30.014) | 21.100 (29.765) | 26.183 (21.945) | 43.617 (41.759)
  2 h | 9.850 (12.188) | 14.633 (25.117) | 35.400 (51.819) | 49.083 (47.324) | 56.550 (36.542) | 75.967 (58.528)
  3 h | 20.667 (20.704) | 41.400 (46.900) | 69.833 (104.167) | 92.717 (56.432) | 136.850 (76.482) | 171.700 (151.630)
  4 h: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
  4 h | 27.180 (21.812) | 57.517 (56.493) | 75.600 (105.466) | 119.183 (24.982) | 192.900 (141.040) | 253.817 (193.963)
  6 h: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
  6 h | 26.060 (12.777) | 55.283 (39.530) | 94.133 (80.855) | 269.000 (108.030) | 193.167 (96.837) | 289.000 (161.294)
  8 h: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
  8 h | 19.640 (9.588) | 41.983 (32.838) | 64.300 (62.242) | 331.500 (167.240) | 128.033 (46.099) | 225.083 (157.281)
  10 h: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 6
  10 h | 29.500 (23.021) | 42.850 (25.960) | 49.533 (57.750) | 253.200 (128.657) | 98.183 (40.408) | 184.950 (138.262)
  12 h: number analyzed (Participants) | 2 | 3 | 5 | 6 | 6 | 6
  12 h | 24.650 (12.657) | 40.267 (19.204) | 41.160 (46.266) | 213.317 (107.529) | 70.817 (13.916) | 142.133 (111.611)
  14 h: number analyzed (Participants) | 2 | 3 | 3 | 6 | 6 | 6
  14 h | 19.550 (7.000) | 30.733 (12.834) | 45.833 (46.048) | 157.517 (89.539) | 54.467 (12.268) | 105.583 (85.266)
  24 h: number analyzed (Participants) | 1 | 3 | 2 | 6 | 6 | 6
  24 h | 12.500 | 20.200 (6.920) | 45.850 (50.558) | 68.417 (34.600) | 38.833 (12.325) | 74.917 (88.938)
  36 h: number analyzed (Participants) | 0 | 3 | 1 | 5 | 6 | 6
  36 h |  | 16.900 (3.672) | 53.600 | 49.340 (20.900) | 35.933 (6.907) | 63.617 (78.709)
  48 h: number analyzed (Participants) | 0 | 3 | 1 | 5 | 3 | 4
  48 h |  | 12.533 (1.704) | 48.500 | 35.720 (13.997) | 29.333 (9.868) | 76.200 (89.700)
  60 h: number analyzed (Participants) | 0 | 2 | 1 | 5 | 3 | 3
  60 h |  | 12.750 (0.919) | 34.900 | 32.500 (13.927) | 25.467 (9.382) | 99.667 (93.713)
  72 h: number analyzed (Participants) | 0 | 0 | 1 | 4 | 5 | 2
  72 h |  |  | 32.100 | 34.175 (8.730) | 25.860 (11.428) | 114.550 (77.004)
  144 h: number analyzed (Participants) | 0 | 0 | 1 | 3 | 3 | 2
  144 h |  |  | 13.800 | 23.167 (2.901) | 12.833 (2.113) | 48.300 (17.112)
  312 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  480 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: VT-11134 Concentrations in Plasma
Description: Mean and standard deviation of VT-11134 concentrations in plasma by nominal time point.
Time Frame: 0 h, 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 14 h, 24 h, 36 h, 48 h, 60 h, 72 h, 144 h, 312 h, and 480 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL
  0 h | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  0.5 h | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.173 (0.425) | 0.000 (0.000) | 0.000 (0.000)
  1 h | 0.185 (0.453) | 0.000 (0.000) | 1.360 (2.692) | 2.320 (3.618) | 2.462 (3.858) | 5.213 (4.512)
  1.5 h | 2.363 (1.972) | 0.417 (0.662) | 7.052 (13.110) | 12.870 (19.273) | 10.290 (9.801) | 18.927 (12.740)
  2 h | 8.763 (6.556) | 1.575 (1.908) | 13.660 (23.209) | 25.947 (33.194) | 24.652 (18.888) | 31.732 (17.109)
  3 h | 21.508 (14.538) | 9.078 (8.322) | 25.530 (31.367) | 53.317 (52.224) | 54.845 (35.132) | 65.550 (31.354)
  4 h | 25.748 (16.413) | 17.412 (10.501) | 29.200 (21.290) | 65.700 (49.461) | 67.117 (40.162) | 86.100 (27.404)
  6 h | 25.550 (11.905) | 28.478 (13.949) | 46.750 (19.144) | 88.200 (36.162) | 71.200 (35.140) | 114.817 (60.895)
  8 h | 16.617 (6.486) | 21.208 (11.449) | 35.183 (15.010) | 97.317 (34.864) | 52.767 (24.493) | 85.283 (42.353)
  10 h | 15.968 (6.143) | 18.990 (9.337) | 27.117 (9.603) | 86.350 (40.901) | 45.200 (19.940) | 78.183 (33.756)
  12 h | 13.252 (4.307) | 16.015 (8.096) | 21.950 (8.474) | 79.083 (29.108) | 37.167 (17.016) | 60.850 (24.612)
  14 h | 11.377 (4.804) | 12.373 (5.510) | 19.017 (5.872) | 61.433 (18.151) | 30.800 (14.162) | 45.767 (17.898)
  24 h | 8.815 (2.712) | 8.382 (2.757) | 12.680 (3.804) | 35.450 (8.349) | 24.065 (10.721) | 34.950 (7.795)
  36 h | 6.910 (1.674) | 7.332 (2.520) | 12.468 (3.626) | 28.883 (8.619) | 22.122 (9.507) | 31.183 (8.235)
  48 h | 5.872 (1.676) | 5.875 (1.974) | 10.290 (3.267) | 22.833 (5.984) | 15.913 (7.928) | 27.017 (5.527)
  60 h | 6.208 (1.839) | 6.848 (2.578) | 10.890 (3.103) | 21.933 (5.385) | 17.750 (8.877) | 26.583 (4.522)
  72 h | 5.060 (1.682) | 5.580 (2.248) | 8.773 (2.048) | 18.650 (4.542) | 17.125 (5.810) | 22.550 (5.990)
  144 h | 3.817 (1.536) | 3.912 (1.301) | 6.575 (2.863) | 15.067 (2.522) | 11.732 (3.208) | 17.583 (5.711)
  312 h: number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 6
  312 h | 2.030 (0.433) | 3.138 (1.902) | 2.965 (1.575) | 9.965 (4.478) | 7.183 (2.189) | 9.357 (6.828)
  480 h: number analyzed (Participants) | 0 | 2 | 2 | 5 | 5 | 6
  480 h |  | 2.010 (0.368) | 3.010 (0.636) | 5.974 (3.631) | 3.982 (2.234) | 4.122 (4.557)

10. Secondary Outcome: Maximum Observed Concentration (Cmax) of VT-1598 and VT-11134
Description: Mean and standard deviation (SD) of the Cmax (ng/mL) PK parameter was estimated from the VT-1598 and VT-11134 plasma concentration-time data.
Time Frame: 0 h through 480 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL
  VT-1598 | 35.43 (17.97) | 63.93 (50.38) | 108.1 (95.57) | 351.0 (148.9) | 222.2 (121.4) | 322.3 (188.4)
  VT-11134 | 30.05 (13.47) | 28.51 (13.89) | 51.02 (25.09) | 108.3 (44.81) | 73.63 (37.55) | 118.6 (57.53)

11. Secondary Outcome: Dose-normalized Maximum Observed Concentration (Cmax/Dose) of VT-1598 and VT-11134
Description: Mean and standard deviation (SD) of the dose-normalized Cmax (ng/mL) PK parameter was estimated from the VT-1598 and VT-11134 plasma concentration-time data.
Time Frame: 0 h through 480 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: (ng/mL)/mg
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
(ng/mL)/mg
  VT-1598 | 0.8858 (0.4492) | 0.7992 (0.6298) | 0.6756 (0.5973) | 2.194 (0.9307) | 0.6943 (0.3793) | 0.5036 (0.2945)
  VT-11134 | 0.7513 (0.3368) | 0.3564 (0.1737) | 0.3189 (0.1568) | 0.6769 (0.2800) | 0.2301 (0.1173) | 0.1853 (0.08989)

12. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of VT-1598 and VT-11134
Description: Mean and standard deviation (SD) of the Tmax (h) PK parameter was estimated from the VT-1598 and VT-11134 plasma concentration-time data.
Time Frame: 0 h through 480 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
h
  VT-1598 | 5.00 (2.68) | 5.00 (1.10) | 4.83 (1.33) | 8.17 (3.49) | 5.05 (1.05) | 4.83 (1.33)
  VT-11134 | 5.50 (2.51) | 5.67 (0.818) | 5.17 (1.33) | 7.67 (2.94) | 5.05 (1.05) | 6.33 (1.97)

13. Secondary Outcome: Terminal Elimination Half-life (t 1/2) of VT-1598 and VT-11134
Description: Mean and standard deviation (SD) of the t 1/2 (h) PK parameter was estimated from the VT-1598 and VT-11134 plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 2.0 half-lives, and includes at least 3 timepoints after Tmax.
Time Frame: 0 h through 480 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 3 | 3 | 5 | 6 | 6 | 6
h
  VT-1598 | 5.403 (3.233) | 29.07 (11.31) | 17.11 (25.09) | 61.38 (54.52) | 40.70 (16.36) | 33.57 (31.79)
  VT-11134 | 117.8 (50.49) | 181.7 (127.9) | 158.5 (90.62) | 249.3 (177.2) | 272.0 (174.7) | 210.7 (217.2)

14. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Concentration Above the Lower Limit of Quantification (AUC(0-last)) of VT-1598 and VT-11134
Description: Mean and standard deviation (SD) of the AUC(0-last) (h*ng/mL) PK parameter was estimated from the VT-1598 and VT-11134 plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 2.0 half-lives, and includes at least 3 timepoints after Tmax.
Time Frame: 0 h through 480 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL
  VT-1598 | 214.2 (183.9) | 894.3 (793.1) | 1540 (2726) | 6293 (3229) | 4177 (1643) | 7730 (9144)
  VT-11134 | 1233 (500.7) | 1551 (628.5) | 2560 (857.3) | 6838 (1459) | 5375 (1513) | 7342 (1866)

15. Secondary Outcome: Dose-normalized Area Under the Concentration-time Curve From Time Zero to the Last Concentration Above the Lower Limit of Quantification (AUC(0-last)) of VT-1598 and VT-11134
Description: Mean and standard deviation (SD) of the dose-normalized AUC(0-last) (h*ng/mL) PK parameter was estimated from the VT-1598 and VT-11134 plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 2.0 half-lives, and includes at least 3 timepoints after Tmax.
Time Frame: 0 h through 480 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: (h*ng/mL)/mg
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
(h*ng/mL)/mg
  VT-1598 | 5.354 (4.598) | 11.18 (9.914) | 9.623 (17.04) | 39.33 (20.18) | 13.05 (5.135) | 12.08 (14.29)
  VT-11134 | 30.81 (12.52) | 19.39 (7.856) | 16.00 (5.358) | 42.74 (9.117) | 16.80 (4.727) | 11.47 (2.916)

16. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC(0-inf)) of VT-1598 and VT-11134
Description: Mean and standard deviation (SD) of the AUC(0-inf) (h*ng/mL) PK parameter was estimated from the VT-1598 and VT-11134 plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 2.0 half-lives, and includes at least 3 timepoints after Tmax.
Time Frame: 0 h through 480 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 1 | 0 | 4 | 3 | 3 | 5
h*ng/mL
  VT-1598: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3
  VT-1598 |  |  |  |  | 5445 (2652) | 2797 (515.0)
  VT-11134 | 1960 |  | 3005 (875.4) | 6923 (1046) | 6260 (703.8) | 7506 (2357)

17. Secondary Outcome: Dose-normalized Area Under the Concentration-time Curve From Time Zero to Infinity (AUC(0-inf)) of VT-1598 and VT-11134
Description: Mean and standard deviation (SD) of the dose normalized AUC(0-inf) (h*ng/mL) PK parameter was estimated from the VT-1598 and VT-11134 plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 2.0 half-lives, and includes at least 3 timepoints after Tmax.
Time Frame: 0 h through 480 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: (h*ng/mL)/mg
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 1 | 0 | 4 | 3 | 3 | 5
(h*ng/mL)/mg
  VT-1598: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3
  VT-1598 |  |  |  |  | 17.02 (8.286) | 4.370 (0.8047)
  VT-11134 | 49.00 |  | 18.78 (5.471) | 43.27 (6.540) | 19.56 (2.199) | 11.73 (3.683)

18. Secondary Outcome: Apparent First-order Elimination Rate Constant (Lambda Z) of VT-1598 and VT-11134
Description: Mean and standard deviation (SD) of the lambda Z (1/h) PK parameter was estimated from the VT-1598 and VT-11134 plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 2.0 half-lives, and includes at least 3 timepoints after Tmax.
Time Frame: 0 h through 480 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 1 | 0 | 4 | 3 | 3 | 5
1/h
  VT-1598: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3
  VT-1598 |  |  |  |  | 0.01940 (0.009617) | 0.06553 (0.03096)
  VT-11134 | 0.005900 |  | 0.006863 (0.001642) | 0.005457 (0.001711) | 0.005520 (0.002165) | 0.006034 (0.001700)

19. Secondary Outcome: Apparent Oral Clearance (CL/F) of VT-1598 and VT-11134
Description: Mean and standard deviation (SD) of the CL/F (L/h) PK parameter was estimated from the VT-1598 and VT-11134 plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 2.0 half-lives, and includes at least 3 timepoints after Tmax.
Time Frame: 0 h through 480 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 1 | 0 | 4 | 3 | 3 | 5
L/h
  VT-1598: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3
  VT-1598 |  |  |  |  | 66.6 (32.4) | 235 (43.8)
  VT-11134 | 20.4 |  | 56.6 (15.6) | 23.5 (3.50) | 51.5 (5.65) | 90.7 (21.8)

20. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vd/F) of VT-1598 and VT-11134
Description: Mean and standard deviation (SD) of the Vd/F (L) PK parameter was estimated from the VT-1598 and VT-11134 plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 2.0 half-lives, and includes at least 3 timepoints after Tmax.
Time Frame: 0 h through 480 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 1 | 0 | 4 | 3 | 3 | 5
L
  VT-1598: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3
  VT-1598 |  |  |  |  | 3440 (28.3) | 4200 (2010)
  VT-11134 | 3460 |  | 8230 (1100) | 4450 (709) | 9410 (922) | 15400 (3820)

21. Secondary Outcome: Cumulative Amount of VT-1598 and VT-11134 Excreted Into Urine From Time Zero to the Time of the Last Quantifiable Concentration (Ae Last)
Description: Mean and (minimum, maximum) of the amount of VT-1598 and VT-11134 excreted into urine from time zero to the time of the last quantifiable concentration.
Time Frame: 0 h through 72 h post dose
Population: as for outcome 8
Measure: Mean (Full Range); unit: mg
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
mg
  VT-1598 | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000]
  VT-11134 | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.00004167 [0.000 to 0.000250] | 0.0008970 [0.000 to 0.00158] | 0.0000 [0.000 to 0.000] | 0.0002200 [0.000 to 0.00132]

22. Secondary Outcome: Percent of VT-1598 Excreted Into Urine (Ae%Dose)
Description: Mean and (minimum, maximum) of the percent of VT-1598 excreted into urine.
Time Frame: 0 h through 72 h post dose
Population: as for outcome 8
Measure: Mean (Full Range); unit: percent
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
percent | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000]

23. Secondary Outcome: Renal Clearance (CLr) of VT-1598 and VT-11134
Description: Mean and standard deviation (SD) of CLr (mL/min) of VT-1598 and VT-11134.
Time Frame: 0 h through 72 h post dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
mL/min
  VT-1598: number analyzed (Participants) | 3 | 3 | 5 | 6 | 6 | 6
  VT-1598 | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  VT-11134 | 0.000 (0.000) | 0.000 (0.000) | 0.000460 (0.00113) | 0.00510 (0.00338) | 0.000 (0.000) | 0.000957 (0.00234)

ADVERSE EVENTS:
Time Frame: Day 1 (ingestion of study product) through Day 21
Description: Any medical or laboratory condition present at the time of screening up through ingestion of the dose was considered as baseline/pre-existing condition and was not reported as an AE. If the severity of any condition increased at any time during the study after ingestion of the dose, it was recorded as an AE.
Arm/Group | 40 mg Fasted | 80 mg Fasted | 160 mg Fasted | 160 mg Fed | 320 mg Fasted | 640 mg Fasted | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 5/6 | 3/6 | 5/6 | 11/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 40 mg Fasted (N=6) | 80 mg Fasted (N=6) | 160 mg Fasted (N=6) | 160 mg Fed (N=6) | 320 mg Fasted (N=6) | 640 mg Fasted (N=6) | Placebo (N=12)
Infusion site thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic decreased (Investigations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Heart rate decreased (Investigations) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cortisol decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Basophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 4 (4) | 0 (0) | 2 (2) | 3 (3) | 1 (2) | 3 (3) | 3 (3)
Respiratory rate increased (Investigations) | 4 (4) | 5 (5) | 4 (7) | 2 (3) | 3 (5) | 1 (1) | 4 (4)
Protein total decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT04208321/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT04208321/SAP_001.pdf